CLINICAL TRIAL: NCT06447363
Title: Assessment of Green Dentistry Knowledge, Attitude and Implementation and Its Association With Sociodemographic Factors Among Undergraduate and Postgraduate Dental Students in Cairo University: A Cross Sectional Study.
Brief Title: Assessment of Green Dentistry Knowledge, Attitude and Implementation and Its Association With Sociodemographic Factors Among Dental Professionals in Cairo University.
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, cinderella khalid, Main Researcher, Cairo University
Other Study IDs: Green Dentistry
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Green Dentistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Environmental pollution is one of the serious issues causing global warming. Each and every individual is responsible for this situation and should make an effort and contribute in keeping the planet green and make it a better place to live for future generations. With escalating contamination of natural resources due to mounting waste generation across industries, including healthcare, the global shift towards ecological sustainability becomes imperative.

The aim of this study is to endeavors to evaluate the knowledge, behavior, and implementation of eco-friendly dental strategies among dental professionals (undergraduate and postgraduate dental students) in the Faculty of Dentistry, Cairo University, and its association with sociodemographic data utilizing self-reporting questionnaire in preparation for the implementation of eco-friendly dental practices.

ELIGIBILITY:
Inclusion Criteria:

* Dental professionals (Undergraduate and postgraduate students), Faculty of Dentistry, Cairo University through the academic year 2024-2025.

Exclusion Criteria:

* Dental students from other universities.
* Internship dental students.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Dental professionals (Undergraduate and postgraduate students), Faculty of Dentistry, Cairo University through the academic year 2024-2025.
Sampling Method: Probability Sample
Enrollment: 553 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge | 1 year
  Unit of measurement is Dichotomous (Yes/No)

SECONDARY OUTCOMES:
Attitude and implementation | 1 year
  Unit of measurement is Dichotomous (Yes/No)